CLINICAL TRIAL: NCT01561001
Title: 24-hour Intraocular Pressure Fluctuation Profile Recorded With SENSIMED Triggerfish® in Patients With Primary Open Angle Glaucoma Before and After Deep Sclerectomy With Collagen Implant
Brief Title: IOP Fluctuations in Primary Open Angle Glaucoma Patients Before and After Deep Sclerectomy With Collagen Implant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Sensimed AG (Industry)
Collaborators: Clinique Monchoisi (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TF-1113
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: SENSIMED Triggerfish® — Portable investigational device using a contact lens sensor that monitors the IOP fluctuation continuously over 24-hours.

SUMMARY:
Primary open angle glaucoma (POAG) is associated with inadequate drainage of the aqueous humor via the trabecular meshwork towards the systemic circulation. This may lead to an increase in IOP and may damage the optic nerve. The purpose of glaucoma management is to lower IOP in order to prevent progression of the optic neuropathy and subsequent visual loss. Firstline treatment usually includes IOP-lowering drug therapy. However, if IOP remains uncontrolled and/or the optic nerve damage progresses despite controlled IOP, surgery may be indicated. Deep sclerectomy with a collagen implant (DSCI) is a non-penetrating surgical procedure for the treatment of open angle glaucoma that allows the enhancement of the aqueous outflow. This forms the rationale to conduct this prospective, open label study to assess the 24-hour IOP fluctuation profile recorded with Triggerfish® in patients with POAG before and after DSCI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of POAG
* Documented glaucomatous VF damage with mean defect (MD) > 3 dB
* Progressing glaucomatous damage justifying a DSCI
* Aged ≥18 years, of either sex
* Not more than 4 diopters spherical equivalent on the study eye
* Not more than 2 diopters cylinder equivalent on the study eye
* Have given written informed consent, prior to any investigational procedures

Exclusion Criteria:

* Corneal or conjunctival abnormality precluding contact lens adaptation
* Severe dry eye syndrome
* Patients with allergy to corneal anesthetic
* Patients with contraindications for silicone contact lens wear
* Patients not able to understand the character and individual consequences of the investigation
* Participation in other clinical research within the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-04; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Effect of DSCI on IOP fluctuation profile as recorded by Triggerfish® in patients with POAG. | 3 months
  The IOP fluctuation profile will be recorded by Triggerfish® in patients with POAG
  * before DSCI
  * 3 months after DSCI.

SECONDARY OUTCOMES:
Effect of DSCI on the diurnal and nocturnal IOP fluctuation pattern | 3 months
  Diurnal and nocturnal IOP fluctuation pattern, wake/sleep and sleep/wake Triggerfish® slopes, Timing of Triggerfish® acrophase, Concomitant IOP-lowering topical drug use
Changes in visual field 3 months after DSCI | 3 months
  Change in the visual field
Safety and tolerability | 3 months
  Adverse events and serious adverse events collected throughout the duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: André Mermoud, MD, Principal Investigator — Clinique Monchoisi, Unité du Glaucome
Locations (1):
- Clinique Monchoisi, Unité du Glaucome, Lausanne, Switzerland